CLINICAL TRIAL: NCT00685321
Title: A Double Blind Randomized Controlled Trial to Explore the Tolerability, Safety and Efficacy of the H-Coil Deep Transcranial Magnetic Stimulation (TMS) in Subjects With Negative Symptoms and Cognitive Deficits of Schizophrenia
Brief Title: Tolerability, Safety and Efficacy of the H1-coil Deep Transcranial Magnetic Stimulation in Subjects With Negative Symptoms and Cognitive Deficits of Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0024-07-SHA
Record Dates: First submitted 2008-05-25; First posted 2008-05-28 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Schizophrenia
Keywords: schizophrenia; TMS; brain stimulation; negative symptoms; clinical improvement; cognitive improvement
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): deep TMS treatment
  Interventions: Device: H1 deep TMS coil
- 2 (Sham Comparator): inactive treatment
  Interventions: Device: Sham

INTERVENTIONS:
Device: H1 deep TMS coil — 20 daily deep rTMS treatment
  Arms: 1
Device: Sham — inactive treatment
  Arms: 2

SUMMARY:
Objectives:The purpose of the study is to explore the efficacy and safety of H1-Coil deep brain rTMS in subjects with negative symptoms and cognitive deficits of schizophrenia (deficit syndrome), currently treated with atypical antipsychotics.

Patient Population: The intention is to treat 45 patients diagnosed with schizophrenia, who are currently suffering mainly from negative symptoms and cognitive deficits (deficit syndrome). The patients will be of all racial, ethnic and gender categories, ranging from 18 to 65 years of age, and have PANSS negative≥21 and PANSS positive<24. Patients will be recruited from both academic and private research centers.

Structure: The study is a randomized, prospective, 8 weeks, double blind study. Blinding: The treatment administrator and the study personnel and patients will be masked to the treatment being administrated.

Concurrent Control: The study group will receive active rTMS treatment and the control group will receive an inactive, sham treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18-65 (male and female), Diagnosed in the past as suffering from schizophrenia. The diagnosis will be reaffirmed according to ICD criteria.
2. Right hand dominant.
3. Scores in PANSS negative questionnaire above 21.
4. Gave informed consent for participation in the study.
5. Negative answers on safety screening questionnaire for transcranial magnetic stimulation
6. stable on the same antipsychotic medication for at least two months prior to entering the study.
7. Negative answers to all questions in the TMS safety questionnaire (attached ).

Exclusion Criteria:

1. Diagnosed as suffering from another axis 1 disorder .
2. Scores in PANSS positive questionnaire above 24.
3. History of epilepsy, seizure, or hot spasm.
4. History of epilepsy within first-degree relatives.
5. History of head injuries.
6. History of metal in the head (outside the mouth space).
7. History of surgery including metal implant or history of metal particles in the eye, pacemaker, or any other medical pump.
8. History of migraines.
9. History of hearing loss (not due to aging) or cochlear implants.
10. History of drug or alcohol abuse during the last year.
11. Women - Pregnancy or not using a reliable method of birth control.
12. Inability to achieve satisfying level of communication with the subject.
13. suicide attempt in the year prior to treatment or suicide risk according to a suicide questionnaire
14. Custodians.
15. Participation in another medical study during the experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-06; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
SANS | 1.5 year

SECONDARY OUTCOMES:
SOFAS | 1.5 Year

CONTACTS AND LOCATIONS:
Overall Officials: yechiel levkovitz, MD, Principal Investigator — Shalvate mental health center
Locations (2):
- Israel (2):
  - Shalvata Mental Helath Center, Hod HaSharon
  - Shalvata, Hod HaSharon